CLINICAL TRIAL: NCT05848986
Title: Study if the Presence of Functional FcERI/RII on the Surface of Human Blood Platelet
Acronym: FERIplaq
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8947
Record Dates: First submitted 2023-03-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-03

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Whole blood, platelet rich plasma Obtained from a constituted biocollection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Flow cytometry — Analysis of blood samples from a health sample's allergic patients and analysis with flow cytometry

SUMMARY:
Anaphylactic shock is the most severe expression of immediate hypersensitivity reactions. The mechanisms leading to these reactions are still poorly understood and may involve platelets, especially in the most severe forms.

The IgE ( ImmunoglobulineE)-mediated mechanism, involving the FcERI(the high-affinity receptor for the Fc region of immunoglobulin E (IgE) receptor present on the surface of mast cells and basophilic cells, is the most common mechanism. The receptors FcERI and FcERII are also described as being present on the surface of blood platelets, which would imply their activation along with the other cells involved. However, studies showing the presence of the FcERI/RII receptors on blood platelets suffer from many biases.

The main objective of the research is to study whether the FcERI/RII receptors are present and functional on the surface of blood platelets from allergic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years-old
* With a protein/drug allergy (hymenoptera, arachide, amoxicillin)
* Confirmed by skin tests and/or challenge test
* With specific IgEs

Exclusion Criteria:

* Patients who refuse to participate to this study
* Patients unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients assessed in the allergy clinic of the Strasbourg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Presence of functionnal FcERI/RII receptors on the surface of blood platelets from allergic patients | 1 day
  After confirmation of the allergy by a well conducted allergy workup

CONTACTS AND LOCATIONS:
Overall Officials: CHARLES AMBROISE TACQUARD, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Les Hôpitaux Universitaires, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No